CLINICAL TRIAL: NCT02202863
Title: Study on the Effects of Wine Grape Pomace Flour, Used as a Dietary Supplement to Increase the Intake of Dietary Fiber and Antioxidants in Human, on Components of Metabolic Syndrome, Plasma Antioxidants, Oxidative Stress Markers and Inflammatory Markers
Brief Title: Effects of Wine Grape Pomace Flour Used as a Dietary Supplement on Metabolic Syndrome Components
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-029; FONDEF AF10 I1014 (Other: CONICYT CHILE)
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Metabolic Syndrome X; Oxidative Stress
Keywords: Dietary intervention; Wine grape pomace flour; Metabolic Syndrome; Oxidative stress; Antioxidants; Fiber
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Red Wine Grape Pomace Flour (WGPF) (Experimental): Subjects were asked to maintain their regular eating habits and lifestyles for 16 weeks, except for the daily intake of 20 g of WGPF. WGPF was consumed in bread, biscuits or as flour mixed with water during lunch. Bread and biscuits with 20% WGPF were prepared especially in a bakery. WGPF intake was supervised every day at lunch. Participants were asked to consume the flour supplement with their regular meals on weekends.
  Interventions: Dietary Supplement: Red wine grape pomace flour (WGPF)
- Control (No Intervention): Subjects were asked to maintain their regular eating habits and lifestyles for 16 weeks.

INTERVENTIONS:
Dietary Supplement: Red wine grape pomace flour (WGPF) — Pomace, a byproduct from wine production, was obtained from red wine grapes, Cabernet Sauvignon, vintage 2011, Maipo Valley, Chile, after alcoholic fermentation. The wine grape pomace was dried and grounded to obtain the flour. Intervention group ate 20 g per day of this flour, which contained 10 g of dietary fiber and an antioxidant capacity of 7,258 ORAC units.
  Arms: Red Wine Grape Pomace Flour (WGPF)

SUMMARY:
Lifestyle modifications, including healthy food intake, exercise, and suppression of tobacco smoking, constitute the most powerful tool to fight chronic diseases. Antioxidants and fiber, two components of Mediterranean diets, are key functional elements for healthy eating and nutrition. We prepared flour from wine grape pomace (WGPF), a rich source of antioxidant and fiber, to be used as an ingredient for functional foods and as a dietary supplement to increase the intake of dietary fiber and bioactive compounds. WGPF was obtained from red grapes (Cabernet Sauvignon variety, Chile). The byproduct of pressing crushed grapes after alcoholic fermentation was dried, grounded and stored. The purpose of this study is to determine the effects of red wine grape pomace flour intake on glycaemia, plasma lipid profile, plasma antioxidants (vitamin C and E), oxidative stress and inflammatory markers.

DETAILED DESCRIPTION:
A 16-week longitudinal intervention study. Males, 30-65 years of age, with at least one component of metabolic syndrome, were randomly assigned to either the intervention group or the control group. At lunch, the intervention group was given 20 g of WGPF per day, which contained 10 g of dietary fiber and an antioxidant capacity of 7,258 ORAC (oxygen radical absorbance capacity) units. Both groups were asked to maintain their regular eating habits and lifestyles. Clinical evaluation, anthropometric measurements and biochemical blood analyses were done at the beginning and the end of the study.

The intervention was carried out at a heavy mining machinery company in Santiago, Chile. All employees were informed about the study and invited to participate. Initially, 47 male workers free of exclusion criteria agreed to participate. The number of participants in each group was chosen based on the variation coefficients in the evolution of total cholesterol in the intervention and in the control group, observed in a previous work (Jiménez, J.P., et al., Effects of grape antioxidant dietary fiber in cardiovascular disease risk factors. Nutrition, 2008. 24(7-8): 646-53).

Statistical analysis: Continuous variables will be shown as mean and standard deviation, while categorical variables as the number of cases and percentage. The student t-test for independent samples and the chi-square test will be used to analyze differences of means and proportions between the two groups, respectively. The student t-test for paired samples and McNemar's test will be used to analyze differences of means and proportions within each group. When appropriate, the Wilcoxon signed rank-sum test will be used to compare paired medians. All p values will be two-tailed and a value <0.05 will be considered to be statistically significant. Data processing and statistical analyses will be done with the SAS statistical software package version 9.1 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Subject who regularly consumed an omnivorous diet.
* Subjects that had at least one of the five components of metabolic syndrome.

Exclusion Criteria:

* Subjects that were under treatment for diabetes mellitus, hypertension (> 160/100) or dyslipidemia (hypertriglyceridemia> 500 mg / dl, hypercholesterolemia> 350 mg / dl)
* Subjects who consume drugs affecting lipid profile, blood pressure, metabolism of carbohydrates or the antioxidant capacity of plasma.
* Subjects with obesity, BMI > 30
* Subjects who have had a cardiovascular event.
* Subjects with bariatric surgery
* Subjects with untreated thyroid disease, renal disease (serum creatinine> 1.5 mg / dl), active liver disease, or other rheumatic disease that could alter the measurements.
* Subjects with chronic inflammatory diseases.
* Subjects that use of supplements containing antioxidants.
* Smoking more than 5 cigarettes per day

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Metabolic Syndrome | Baseline and 16 weeks
  The presence of metabolic syndrome components was defined using the criteria proposed by the Adult Treatment Panel III of the US National Cholesterol Education Program: (i) abdominal obesity as waist circumference >102 cm for men; (ii) low levels (<40 mg/dL for men) of serum high density lipoprotein cholesterol; (iii) hypertriglyceridemia as 150 mg/dL or more; (iv) elevated blood pressure as 130/85 mm Hg or higher; and (v) impaired glucose homeostasis as fasting plasma glucose levels of 100 mg/dL or higher

SECONDARY OUTCOMES:
Postprandial insulin | Baseline and 16 weeks
  An oral glucose tolerance test (OGTT) was performed after overnight fasting. Subjects ingested a solution containing 75 g of dextrose, and venous blood samples were obtained at 0 and 120 min to determine plasma glucose and insulin levels. Insulin was measured by electrochemiluminescence immunoassay (ECLIA; Roche Diagnostics®).

OTHER OUTCOMES:
Antioxidants | Baseline and 16 weeks
  Antioxidants measurements: Total Plasma Antioxidant Capacity (TRAP), Total Plasma Antioxidant Reactivity (TAR), Vitamin C and Vitamin E.
Oxidative stress | Baseline and 16 weeks
  Oxitative stress markers: Malondialdehyde (MDA), Protein Carbonyl and the Methionine Sulfoxide in plasma.
Inflammation | Baseline and 16 weeks
  Inflammatory markers: Tumor Necrosis Factor -Alfa, IL-6, Monocyte Chemotactic Protein -1, in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Ines Urquiaga, Ph.D, Principal Investigator — Centro de Nutricion y Enfermedades Cronicas, Pontificia Universidad Catolica de Chile
Locations (1):
- Centro de Nutricion Molecular y Enfermedades Cronicas, Pontificia Universidad Catolica de Chile, Santiago, Centro, Chile